CLINICAL TRIAL: NCT04095572
Title: Non-antimicrobial Alternative in Prophylaxis of Recurrent Urinary Tract Infections: a Prospective, Randomised-controlled, Double-blinded, Multicentre Study
Brief Title: Alternative Prophylaxis in Female Recurrent Urinary Tract Infections
Acronym: AlP-FrUiT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-01377; me19Bausch
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Urinary Tract Infections; Urinary Tract Infection (UTI)
Keywords: Hyaluronic acid (HA); Chondroitin sulphate (CS); antimicrobial resistance rates; Intravesical instillation; HA-CS instillations; Recurrent Urinary Tract Infection (rUTI)
MeSH Terms: conditions — Urinary Tract Infections | interventions — Administration, Intravesical

STUDY DESIGN:
Intervention Model Description: Pragmatic, parallel arm, superiority, multicentre, randomised trial with blinded treating physicians, patients and outcome assessors
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group A (Active Comparator): 50 ml of a sterile sodium HA (800 mg)- CS (1g) solution (Ialuril Prefill®, IBSA Farmaceutici Italia Srl, Via Martiri di Cefalonia 2, 26900 Lodi, Italy) weekly for four weeks, then every second week in the second month and four weeks later
  Interventions: Drug: intravesical instillation with HA-CS
- control group B (Placebo Comparator): 50 ml sterile purified water weekly for four weeks, then every second week in the second month and four weeks later
  Interventions: Drug: intravesical instillation of sterile purified water

INTERVENTIONS:
Drug: intravesical instillation with HA-CS — intravesical instillation with HA-CS (Ialuril Prefill®, IBSA Farmaceutici Italia Srl, Lodi, Italy)
  Arms: intervention group A
Drug: intravesical instillation of sterile purified water — intravesical instillation of sterile purified water (packed and labelled according to Good Manufacturing Practice at IBSA Farmaceutici Italia Srl in Lodi, Italy to provide adequate blinding)
  Arms: control group B

SUMMARY:
Urological pathogens are effected by rising antimicrobial resistance rates due to the frequent use of antimicrobials for treatment and prophylaxis. Intravesical instillation with hyaluronic acid (HA) and chondroitin sulphate (CS) obtained positive outcomes in the treatment of overactive bladder, radiation cystitis and interstitial cystitis by replenishment of the glycosaminoglycan layer of the bladder. This study is to investigate whether intravesical instillation with HA-CS in patients with recurrent urinary tract infections (rUTI) is superior to a placebo instillation in terms of reduction of rate of symptomatic urinary tract infections (UTIs) (based on clinical diagnosis) needing treatment with antimicrobials within 12 months after randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of rUTI, defined as ≥ 3 episodes of (un)complicated UTI documented by urine culture with the isolation of ≥103 cfu/ml of an identified pathogen in the last year with clinical symptoms OR 2 episodes in the last 6 month

Exclusion Criteria:

* No informed consent
* Concomitant UTI (< 7 days prior to randomisation)
* Ongoing antimicrobial prophylaxis (e.g. for rUTI or for any other reason like endocarditis, transplanted patients under immunosuppression)
* Ongoing prophylactic strategy (e.g. immunoactive prophylaxis)
* Documented underlying urogenital abnormality (e.g. significant post voiding residual volume (>50 ml), urethral stricture, urethral diverticula, urinary stone, reflux, urinary neoplasia), urological device (e.g. catheter, ureteral stent) or symptomatic pelvic floor disorder (e.g. genital prolapse stage ≥ II)
* Concomitant disease (i.e. renal insufficiency, diabetes mellitus, corticosteroid use)
* Urogenital urological or gynecological surgery < 6 weeks
* Known allergy to the study medication
* Use of spermicides or intrauterine device
* Pregnancy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of symptomatic UTIs (based on clinical diagnosis) needing treatment with antimicrobials | within 12 months after randomisation
  Rate of symptomatic UTIs (based on clinical diagnosis) needing treatment with antimicrobials (cumulative number)

SECONDARY OUTCOMES:
Symptomatic UTI (based on clinical diagnosis supported by measured bacteriuria of ≥103 cfu/ml) treated with antimicrobials | at screening and at each instillation visit (week 1 = Randomization, week 2, week 3, week 4, week 6, week 8, week 12) and at follow-up visits after randomization (month 6, month 9, month 12)
  Symptomatic UTI (based on clinical diagnosis supported by measured bacteriuria of ≥103 cfu/ml) treated with antimicrobials (cumulative number)
Symptoms of UTI according to the Acute Cystitis Symptom Score (ACSS) (cumulative number of each symptom) | at screening and at each instillation visit (week 1 = Randomization, week 2, week 3, week 4, week 6, week 8, week 12) and at follow-up visits after randomization (month 6, month 9, month 12)
  Change in Acute Cystitis Symptom Score (ACSS). The first part of the ACSS questionnaire consists of 14 questions. The first 6 questions assess typical symptoms of UTI: frequency, urgency, pain and burning during urination, sensation of incomplete bladder emptying, pain/discomfort in the lower abdomen, visible hematuria. Each question concerning urinary symptoms allows the patient to choose one out of four answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 3. The score can range between 0 and 18. It has been validated and a score ≥ 6 seems to be very indicative for the diagnosis of an UTI.
Time to UTI recurrence (as days between randomisation and the first recurring UTI) | at screening and at each instillation visit (week 1 = Randomization, week 2, week 3, week 4, week 6, week 8, week 12) and at follow-up visits after randomization (month 6, month 9, month 12)
  Time to UTI recurrence (as days between randomisation and the first recurring UTI)
Asymptomatic bacteriuria of ≥105 cfu/ml | at each instillation visit (week 1 = Randomization, week 2, week 3, week 4, week 6, week 8) if the urine dipstick is suspicious, at the 7th instillation (= week 12 )and at 12 month follow-up
  Asymptomatic bacteriuria, measured by number of colony forming Units (cfu) of ≥105 cfu/ml
Detection of multidrug-resistant bacteria in urine culture (3Multiresistant gram negatives (MRGN), 4MRGN) | at screening and at at each instillation visit (week 1 = Randomization, week 2, week 3, week 4, week 6, week 8, week 12) and at follow-up visits after randomization (month 6, month 9, month 12)
  Detection of multidrug-resistant bacteria in urine culture (3MRGN, 4MRGN) (yes/no)
Prescribed defined daily doses (DDD) of antibiotics (cumulative sum of DDD) | from randomisation to 12 months
  Prescribed defined daily doses (DDD) of antibiotics (cumulative sum of DDD)
Change in Pelvic Pain and Urinary/Frequency (PUF) Symptom Scale | prior to randomisation and at 1 month, 3 months, 6 months, 9 months, 12 months
  The PUF questionnaire consists of 12 questions. The first two questions allow the patient to choose one out of five answers (points 0-3), the following questions one out of four (points 0-3) indicating increasing severity of the particular symptom. Seven of the questions concern symptoms (total count 23), four questions are part of the bother score (total count 12). Total score consists of symptom score and bother score (total count 35). The change of the score is calculated by subtracting the score at 1 month, 3 months, 6 months, 9 months, 12 months from the score at enrolment
Change in QoL Short Form (SF)-36 score | prior to randomisation and at 12 months
  The QoL SF-36 consists of 36 items including eight independent scales and two main dimensions 35 of the items are compressed into eight multi-item scales: (1) physical functioning is a ten-question scale; (2) role-physical is a four-item scale; (3) bodily pain is a two-item scale; (4) general health is a five-item scale; (5) vitality is a four-item scale; (6) social functioning is a two-item scale; (7) role-emotional is a three-item scale; and (8) mental health is a five-item scale. Hence, in the SF-36 scoring system, the scales are assessed quantitatively, each on the basis of answers to two to ten multiple choice questions, and a score between 0 and 100 is then calculated on the basis of well-defined guidelines, with a higher score indicating a better state of health. The change of the score is calculated by subtracting the score at 12 month from the score at enrolment.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Bausch, Dr. med, Principal Investigator — Department of Urology, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Department of Gynecology, University Hospital Basel, Basel
  - Department of Urology, University Hospital Basel, Basel